CLINICAL TRIAL: NCT03104790
Title: Assessment of Viral Shedding in Children Previously in Receipt of Multiple Doses of Live Attenuated Influenza Vaccine (LAIV) Compared to Influenza Vaccine-naïve Controls
Acronym: Flushed
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Flushed
Record Dates: First submitted 2017-03-23; First posted 2017-04-07 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-04

CONDITIONS: Influenza Vaccination; Influenza; Vaccination
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Two groups based on prior vaccination history
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- naive (Experimental): Children who have never received any influenza vaccine (The two groups are defined by immunisation history, all receive the same intervention in the study)
  Interventions: Biological: Fluenz Tetra (The two groups are defined by immunisation history, all receive the same intervention in the study)
- prior vaccinees (Experimental): Children who have received at least two doses of Fluenz Tetra previously (The two groups are defined by immunisation history, all receive the same intervention in the study)
  Interventions: Biological: Fluenz Tetra (The two groups are defined by immunisation history, all receive the same intervention in the study)

INTERVENTIONS:
Biological: Fluenz Tetra (The two groups are defined by immunisation history, all receive the same intervention in the study) — live attenuated influenza vaccine (LAIV)

SUMMARY:
LAIV shedding studies in children could be an important way to confirm whether impediments to viral replication do indeed explain these observed reductions in vaccine effectiveness(VE), whether prior vaccination has any influence on replication and what future implications (if any) this might have for the UK paediatric LAIV programme. LAIV virus replication in children will be dependent on virological and host factors. The virus factors include replicative fitness of individual strains and the susceptibility to inhibition by other replicating strains (ability to compete). Host factors which may influence this include pre-existing specific immunity as a result of prior infection or previous vaccination (with either LAIV or IIV), and innate immune factors including mucosal immunity. Understanding the relative importance of different factors over two seasons when the strain composition of the A/H1N1pdm09 LAIV virus will change and by comparing previously unvaccinated and highly vaccinated groups (with both LAIV and IIV), can potentially give unique insights into their contribution to the US LAIV observations.

With the change of the A/H1N1pdm09 vaccine strain in 2017/18, demonstrating improved performance (in terms of VE, virus shedding and immunogenicity) and what contribution prior vaccination might make will be key evidence for both the UK, but also the US. Information presented at the ACIP in June 2018 from the 2016/17 and 2017/18 seasons will be key to inform US future decisions around use of LAIV.

This is a parallel group, non randomised study which will enrol at least 400 children. Both written informed consent from parent/ guardian and written assent from the child will be in place prior to any study procedure. The two groups will be defined by previous influenza vaccination history, with around half the children naïve to any influenza vaccination (LAIV or IIV) and half having had at least three doses of LAIV with or without IIV. All will follow the same schedule of vaccination and oral fluid collection at day 0 (by the nurse in the home or at the GP surgery); nasal swab collection (by the parent at home on days 1,3,6); day 21 oral fluid collection (by nurse or parent at home or at GP surgery).

DETAILED DESCRIPTION:
The United States of America (USA) has a long-standing paediatric influenza vaccination programme, including use of live attenuated influenza vaccine (LAIV). Following evidence of lack effectiveness of LAIV in 2015/16, the USA suspended use in the 2016/17 season. The UK introduced LAIV for children in 2013/14 and has since been closely monitoring programme performance. In 2015/16, the UK - in contrast to the USA - found evidence of significant effectiveness of LAIV against laboratory confirmed influenza in both primary and secondary care including against A/H1N1pdm09. The UK results concord with those from several other geographical settings, although several studies report relatively lower effectiveness of LAIV against A/H1N1pdm09 infection compared to inactivated influenza vaccine (IIV). The reasons for these apparent differences in effectiveness are currently unclear.

The USA has indicated that for the Advisory Committee on Immunisation Practice (ACIP) to rescind their decision to suspend use of LAIV, they will require an understanding of the likely underlying mechanism for the apparent reduction in LAIV A/H1N1pdm09 vaccine effectiveness (VE) measured in observational studies in the USA and then evidence that the problem has been resolved.

Several hypotheses are emerging to explain the apparent reduction in A/H1N1pdm09 quadrivalent LAIV effectiveness in the USA last season and their discordance with findings elsewhere including the UK together with the possible lower effectiveness of LAIV against A/H1N1pdm09 compared to IIV. These include one or more of the following:

1. Center for Disease Control (CDC)/ Department of Defense (DoD) specific finding - related to chance, methodology, programmatic issues
2. Reduced replicative fitness of the current A/H1N1pdm09 strain.
3. Viral interference/competition between A/H1N1pdm09 vaccine strain and other vaccine viruses in multivalent formulation;
4. Prior vaccination with LAIV or IIV resulting in specific immunological interference with H1N1pdm09 vaccine virus replication;
5. Repeat LAIV vaccination resulting in broader, longer term immunological changes affecting all viruses (mimicking adult response);
6. Combinations of the above Based upon in vitro studies, the manufacturer of LAIV (MedImmune) have stated that reduced replicative fitness of the A/H1N1pdm09 strain is likely to be the important root cause. However, this factor alone cannot explain the difference in effectiveness observed between the USA and sites elsewhere including the UK. This suggests that there is an important additional factor(s) involved. The US programme has been running for many more years than the UK - and in addition children 6 months to 24 months of age are offered IIV, unlike the UK. These prior vaccine exposures are potential contributory factors.

LAIV shedding studies in children could be an important way to confirm whether impediments to viral replication do indeed explain these observed reductions in VE, whether prior vaccination has any influence on replication and what future implications (if any) this might have for the UK paediatric LAIV programme. LAIV virus replication in children will be dependent on virological and host factors. The virus factors include replicative fitness of individual strains and the susceptibility to inhibition by other replicating strains (ability to compete). Host factors which may influence this include pre-existing specific immunity as a result of prior infection or previous vaccination (with either LAIV or IIV), and innate immune factors including mucosal immunity. Understanding the relative importance of different factors over two seasons when the strain composition of the A/H1N1pdm09 LAIV virus will change and by comparing previously unvaccinated and highly vaccinated groups (with both LAIV and IIV), can potentially give unique insights into their contribution to the US LAIV observations.

With the change of the A/H1N1pdm09 vaccine strain in 2017/18, demonstrating improved performance (in terms of VE, virus shedding and immunogenicity) and what contribution prior vaccination might make will be key evidence for both the UK, but also the US. Information presented at the ACIP in June 2018 from the 2016/17 and 2017/18 seasons will be key to inform US future decisions around use of LAIV.

This is a parallel group, non randomised study which will enrol at least 400 children. Both written informed consent from parent/ guardian and written assent from the child will be in place prior to any study procedure. The two groups will be defined by previous influenza vaccination history, with around half the children naïve to any influenza vaccination (LAIV or IIV) and half having had at least three doses of LAIV with or without IIV. All will follow the same schedule of vaccination and oral fluid collection at day 0 (by the nurse in the home or at the GP surgery); nasal swab collection (by the parent at home on days 1,3,6); day 21 oral fluid collection (by nurse or parent at home or at GP surgery).

ELIGIBILITY:
Inclusion Criteria:

-

Children may only be included in the study if all the inclusion criteria are met:

* Children age 6 to 13 years of age on enrolment and with either:

  * Prior LAIV vaccination in at least 2 out of the 3 previous years
  * Have never received LAIV or IIV in previous years
* Children eligible to receive LAIV in accordance with Green Book advice [https://www.gov.uk/government/organisations/public-health-england/series/immunisation-against-infectious-disease-the-green-book]
* Written informed consent given by parent/ guardian and assent from child (both must be in place to proceed)

Exclusion Criteria:

-

Children may not be included in the study if any of the following apply:

1. Admission to Paediatric ntensice care unit (PICU) for invasive ventilation due to a respiratory illness in the preceding 2 years.
2. Contraindications to LAIV (notwithstanding allergy to egg protein), which include:

   1. Hypersensitivity to the active ingredients, gelatin or gentamicin (a possible trace residue)
   2. Previous systemic allergic reaction to LAIV
   3. Previous allergic reaction to an influenza vaccine (not LAIV) is a relative contra-indication, which must be discussed with the CI to confirm patient suitability
   4. Children/adolescents who are clinically immunodeficient due to conditions or immunosuppressive therapy such as: acute and chronic leukaemias; lymphoma; symptomatic HIV infection; cellular immune deficiencies; and high-dose corticosteroids*.

      *High-dose steroids is defined as a treatment course for at least one month, equivalent to a dose greater than 20mg prednisolone per day (any age), or for children under 20kg, a dose greater than 1mg/kg/day.

      NB: LAIV is not contraindicated for use in individuals with asymptomatic HIV infection; or individuals who are receiving topical/inhaled/low-dose oral systemic corticosteroids or those receiving corticosteroids as replacement therapy, e.g. for adrenal insufficiency.
   5. Children / adolescents younger than 18 years of age receiving salicylate therapy because of the association of Reye's syndrome with salicylates and wild-type influenza infection.
   6. Pregnancy
3. Contraindications to vaccination on that occasion, e.g. due to child being acutely unwell:

   1. Febrile ≥38.0oC in last 72 hours
   2. **Acute wheeze in last 72 hours requiring treatment beyond that normally prescribed for regular use by the child's treating healthcare professional
   3. **Recent admission to hospital in last 2 weeks for acute asthma
   4. **Current oral steroid for asthma exacerbation or course completed within last 2 weeks
   5. Any other significant condition or circumstance which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

      * Items 3b-3d are relative contra-indications: Many children with "difficult-to-control" symptoms fail to meet these criteria on a routine basis. Where these are present, the CI is able to authorise participation on a case-by-case basis, after assessing the child at the time of enrolment.

Administration of another live vaccine (e.g. MMR) within the previous 4 weeks is no longer a contra-indication to LAIV administration, according to updated UK Department of Health guidelines.

NB: See Summary of Product Characteristics for full details of contra-indications to LAIV.

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 373 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
virus shedding | day 0, day 21
  type-specific vaccine virus shedding and immunogenicity in 2017/18 and determine if there has been any change compared to previous studies in 2016/17 (conducted by this group, Eudract 2013-003592-35 and 2016-002352-24) following change in the A/H1N1pdm09 vaccine virus strain amongst children with the same prior vaccine history

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Coates, PhD, Study Chair — Public Health England
Locations (3):
- United Kingdom (3):
  - Gloucestershire primary care, Gloucester, Gloucestershire
  - Hertfordshire primary care, Hertford, Hertfordshire
  - Imperial Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No
not appllicable

REFERENCES:
- [Derived] Jackson D, Pitcher M, Hudson C, Andrews N, Southern J, Ellis J, Hoschler K, Pebody R, Turner PJ, Miller E, Zambon M. Viral Shedding in Recipients of Live Attenuated Influenza Vaccine in the 2016-2017 and 2017-2018 Influenza Seasons in the United Kingdom. Clin Infect Dis. 2020 Jun 10;70(12):2505-2513. doi: 10.1093/cid/ciz719. PMID 31642899